CLINICAL TRIAL: NCT05554640
Title: Clinical Performance of Two Daily Disposable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6495
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the sequence, Test/Control.
  Interventions: Device: Acuvue® Oasys MAX 1-Day; Device: Dailies Total 1
- Control/Test (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the sequence, Test/Control.
  Interventions: Device: Acuvue® Oasys MAX 1-Day; Device: Dailies Total 1

INTERVENTIONS:
Device: Acuvue® Oasys MAX 1-Day — TEST Lens
Device: Dailies Total 1 — CONTROL Lens

SUMMARY:
This is a subject-masked, randomized, bilateral, 2x2 crossover clinical investigation that will assess lens fit acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 40 (inclusive) years of age at the time of screening.
  4. They agree not to participate in other clinical research while enrolled on this study.
  5. They have worn the same brand of soft daily disposable silicone hydrogel contact lenses at least eight hours per day for at least four days per week over the past 4 weeks.
  6. They own a wearable pair of spectacles if needed for distance vision correction (by self-report).
  7. They can attain a best-corrected logMAR distance visual acuity of at least 0.20 in each eye.
  8. They have spherical contact lens prescription in the range -1.00 to -6.00 DS (based on the calculated ocular refraction).
  9. They have up to maximum of 1.00 DC of refractive astigmatism (based on the calculated ocular refraction).

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g., rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study or may pose a risk to study personnel.
  3. They have an ocular disorder which would normally contraindicate contact lens wear.
  4. They have had cataract surgery.
  5. They have had corneal refractive surgery.
  6. They are using any topical medications such as eye drops or ointments.
  7. Any known hypersensitivity or allergic reaction to sodium fluorescein.
  8. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear. See section 9.1 for additional details regarding excluded systemic medications.
  9. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
  10. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  11. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  12. Any Efron Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection), 13. They have a pre-corneal tear film break-up time less than five seconds when evaluated on the DESMD tear film imaging system.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 subjects were enrolled in this study. Of those enrolled, 14 subjects were dispensed at least one study lens, while 2 subjects failed to meet all eligibility criteria. All dispensed subjects completed the study.
Groups:
- Delefilcon A / Senofilcon A: Subjects randomized to receive the delefilcon A lens during period 1 and the senofilcon A lens during period 2.
- Senofilcon A / Delefilcon A: Subjects randomized to receive the senofilcon A lens during period 1 and the delefilcon A lens during period 2.
Period: Period 1
Arm/Group | Delefilcon A / Senofilcon A | Senofilcon A / Delefilcon A
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Delefilcon A / Senofilcon A | Senofilcon A / Delefilcon A
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 4
  Black or African American | 1
  White | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Acceptable Lens Fitting
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope post lens insertion, the 1- and 2-week follow-up evaluations and any unscheduled visits. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The proportion of eyes with acceptable lens fit was reported.
Time Frame: Up to 2-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Groups:
- Delefilcon A: Subjects that wore the delefilcon A lens during either the first or second period of the study.
- Senofilcon A: Subjects that wore the senofilcon A lens in either the first or second period of the study.
Arm/Group | Delefilcon A | Senofilcon A
Number analyzed (Participants) | 14 | 14
Number analyzed (Eyes) | 28 | 28
Proportion of eyes | 100 | 100

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 28 days per subject.
Arm/Group | Delefilcon A | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05554640/Prot_SAP_000.pdf